CLINICAL TRIAL: NCT05328349
Title: Do Psychosocial Factors Predict the Persistence of Shoulder Pain?
Brief Title: Psychosocial Factors of Persistent Shoulder Pain
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Professor, Laval University
Other Study IDs: #2022-2502
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Early Intervention, Educational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Education Program: All participants will have to present shoulder symptoms related to rotator cuff related shoulder pain, which is defined as pain over the deltoid and/or upper arm region, pain associated with arm movement, and familiar pain reproduced with loading or resisted testing during abduction and/or external rotation of the arm.
  Interventions: Behavioral: Education Program

INTERVENTIONS:
Behavioral: Education Program — After the baseline evaluation, all participants will take part in an education intervention, aiming at promoting self-management of shoulder pain, that will include two one-on-one sessions (approximately 30-45 minutes) within 2 weeks with a physiotherapist (1st session right after the baseline evaluation, 2nd session two weeks later). Participants will receive written information regarding shoulder (anatomy and function) and basic pain science and will be directed to watch a series of six educational videos on shoulder pain and function, persistent pain, physical activity, stress, sleep and eating habits. It should be noted that the objective of this study is not to assess the effectiveness of the intervention; the purpose of offering an intervention to participants is to control the intervention that will be received by them.

SUMMARY:
Several studies have shown that in chronic pain conditions, factors such as lack of positivity and resilience, pain catastrophizing, stress, anxiety and depression can contribute to the persistence and maintenance of pain. Thus, the present project will identify psychosocial risk factors that predict the persistence of shoulder pain. Individuals with shoulder pain (n=112) will be recruited. At baseline, the participants will fill a series of questionnaires evaluating different biopsychosocial constructs (resilience, perceived stress, anxiety, depression, pain, disability, pain catastrophizing, self-efficacy, social support, physical activity). After baseline evaluation, the participants will take part in an educational program aimed at promoting self-management of shoulder pain. At the end of the project (6 months), participants will only fill questionnaires evaluating pain and disability. Based on the scores on these questionnaires, the participants will be classified as having persistent shoulder pain or as recovered. Thereafter, statistical analyses will be performed to identify significant predictors for persistent shoulder pain. The primary hypothesis of the study is that low levels of resilience, self-efficacy, social support and physical activity, and high levels of stress, pain, disability, catastrophizing, anxiety and depression will negatively influence the pain response resulting in increased pain ratings and persistent symptoms over time.

DETAILED DESCRIPTION:
A prospective cohort study will be conducted. One hundred and twelve individuals with rotator cuff related shoulder pain (RCRSP) will be evaluated twice: baseline and 6-month after baseline. At baseline, participants will complete a questionnaire on sociodemographic and symptomatology. Then, the participants will be asked to fill questionnaires covering a biopsychosocial spectrum: Brief Resilience Scale (BRS), Perceived Stress Scale (PSS-10), Numeric Pain Rating Scale (NPRS), abbreviated version of the Disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH), Patient-Health Questionnaire - 9 (PHQ-9), General Anxiety Disorder - 7 (GAD-7), Pain Catastrophizing Scale (PCS), Pain Self-Efficacy Questionnaire (PSEQ), Multidimensional Scale of Perceived Social Support (MSPSS) and short version of the International Physical Activity Questionnaire (IPAQ). After the baseline evaluation, participants will take part in an educational program aimed at promoting self-management of shoulder pain. The program will include two one-on-one sessions (approximately 30-45 minutes) within 2 weeks with a physiotherapist. The main reasons to propose an education intervention is that it is usual to receive a rehabilitation intervention when a person presents shoulder pain. It was therefore difficult to expect that the participants would not seek treatment during the study period and therefore that the investigators could only have considered the effect of time (natural evolution of the injury). Finally, at 6-months, participants will only be asked to fill NPRS and QuickDASH. Based on the scores on these questionnaires, the participants will be classified as having persistent shoulder pain or as recovered.The follow-up evaluation will be performed online (6-month follow-up) using RedCap. For the statistical analysis, participants will be dichotomized into 2 subgroups according to whether their symptoms have resolved or not at 6-month, aiming to determine the baseline variables that predict the persistence of pain 6 months after baseline. All variables found to be significant on univariate analyses will be considered potential predictors. Thereafter, logistic regression analyses will be performed to identify significant predictors for persistent rotator cuff related shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, aged between 18 and 60 years old;
2. English or French speakers;
3. Rotator cuff related shoulder pain symptoms - Rotator cuff related shoulder pain diagnosis will be based on the participant history and a clinical assessment performed by an experienced physiotherapist. Participants will have to present shoulder symptoms related to rotator cuff related shoulder pain, which is defined as:

   * pain over the deltoid and/or upper arm region;
   * pain associated with arm movement;
   * familiar pain reproduced with loading or resisted testing during abduction and/or external rotation of the arm.

   Participants will also have to present at least one positive finding in each of the following categories:
   1. painful arc of movement;
   2. positive Neer's or Kennedy-Hawkins Test;
   3. pain on resisted external rotation, resisted abduction or Empty Can Test. A positive cluster of these criteria represents a valid diagnostic cluster;
4. Minimal score of 12 points on the QuickDASH (based on its minimal clinically important difference [MCID]).

Exclusion Criteria:

1. clinical signs of full thickness rotator cuff tears;
2. other shoulder disorders e.g. adhesive capsulitis (restriction of passive glenohumeral movement of at least 25% for 2 or more directions), severe osteoarthritis, fracture, dislocation, severe acromioclavicular joint pathology;
3. previous shoulder surgery;
4. presence of significant co-morbidity e.g. neurological disorders, rheumatoid arthritis;
5. current or past carcinoma;
6. unlikely to be able to perform required clinical assessment tasks or attend the required evaluation and intervention sessions;
7. symptomatic cervical spine pathology, defined as reproduction of symptoms with active physiological cervical spine movements;
8. corticosteroid injection in the last 6 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Potential participants will be recruited from a convenience sample through the electronic mailing lists of Université Laval (>40,000 individuals), social media (mainly Facebook, Twitter and Instagram), the medical communities in Quebec City (advertisements in medical, physiotherapy, radiology clinics and pharmacies) and advertisement with patient advocacy or professional organizations and with unions of workers at risk for rotator cuff related shoulder pain.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
QuickDASH at 6 months | 6 months
  Shoulder pain and function will be evaluated using the abbreviated version of the Disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) questionnaire. The questionnaire consists of 11 items covering 6 domains (daily activities, symptoms, social function, work function, sleep, and confidence) that are scored on a numeric rating scale between 1 (no difficulty) and 5 (unable).
  Participants will be dichotomized into 2 subgroups according to whether their symptoms have resolved or not at 6-month. To do this, the investigators will use the NPRS and QuickDASH scores from the 6-month follow-up. If patients present a score between 0 (no disability) and 11 (minimal clinically important difference - MCID) on the QuickDASH, their symptoms will be considered resolved. Conversely, if their score is greater than 11 on the QuickDASH , their symptoms will be considered unresolved.
NPRS at 6 months | 6 months
  The NPRS will quantify the average pain over the last 7 days. This scale score ranges from 0 (no pain) to 10 (worst pain), and the scale is considered valid and with good reliability to assess individuals with shoulder pain.
  Participants will be dichotomized into 2 subgroups according to whether their symptoms have resolved or not at 6-month. To do this, the investigators will use the NPRS and QuickDASH scores from the 6-month follow-up. If patients present a score between 0 (no disability) and 2 (minimal clinically important difference - MCID) on the NPRS, their symptoms will be considered resolved. Conversely, if their score is greater than 2 on the NPRS, their symptoms will be considered unresolved

SECONDARY OUTCOMES:
QuickDASH at Baseline | Baseline
  Shoulder pain and function will be evaluated using the abbreviated version of the Disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) questionnaire. The questionnaire consists of 11 items covering 6 domains (daily activities, symptoms, social function, work function, sleep, and confidence) that are scored on a numeric rating scale between 1 (no difficulty) and 5 (unable).
NPRS at Baseline | Baseline
  The NPRS will quantify the average pain over the last 7 days. This scale score ranges from 0 (no pain) to 10 (worst pain), and the scale is considered valid and with good reliability to assess individuals with shoulder pain.
Resilience at Baseline | Baseline
  The validated French version of Brief Resilience Scale (BRS) will be used to classify the groups into low or high resilience levels. The BRS aims to measure the individual's ability to recover from a trauma or stress situations. It is composed of 6 items, which negatively or positively assess the stressful situation. Each question presents 5 response options ranging from 1= "strongly disagree" to 5= "strongly agree". Higher scores represent high levels of resilience. Internal consistency of the scale showed Cronbach's alpha of 0.84.
Perceived Stress at Baseline | Baseline
  The Perceived Stress Scale - 10 (PSS-10) translated and adapted to French will be applied to measure the individuals' perceived stress.66 The scale quantifies the extent of how individuals consider stressful situations experienced in the last month. It uses a 10-item scale with a 5-point Likert scale of response (0=never; to 4=always) and higher scores indicate greater perceived stress. The Cronbach alpha for the instrument is 0.83.66
Pain Catastrophizing at Baseline | Baseline
  The Pain Catastrophizing Scale (PCS) translated and validated to French will be used to identify catastrophic thoughts about pain. The PCS is a 13-item scale aiming to quantify pain catastrophizing characterized by magnification, rumination, and helplessness of pain beliefs. Its score ranges from 0 to 52: 0 - best score and 52=worst score, where 52 means higher individual catastrophizing. High internal reliability has been reported in patients with chronic pain with adequate validity and test-retest reliability.
Depressive symptoms at Baseline | Baseline
  The French version of Patient Health Questionnaire-9, a shorter version of the complete PHQ, will be used to self-report depressive symptoms. Each of the nine items can be scored from 0 (not at all) to 3 (nearly every day), and the total scale score ranges from 0-27, where higher scores mean more severity of symptoms. A Cronbach's alpha of 0.86 was demonstrated for the instrument.
Level of Anxiety at Baseline | Baseline
  The French version of the General Anxiety Disorder (GAD-7) will be utilized to evaluate generalized anxiety. Each of the seven items are scored from 0 (not at all) to 3 (nearly every day). The total GAD-7 scale score ranges from 0-21 and higher scores means higher anxiety levels. The scale presents satisfactory internal consistency (Cronbach's alpha=0.89).
Sel-Efficacy at Baseline | Baseline
  The Pain Self-Efficacy Questionnaire (PSEQ) consists of 10 items utilized to measure patient's confidence in performing daily activities despite of pain. Each item is rated on a scale ranging from 0 ("not at all confident") to 6 ("completely confident"), and the total score can range from 0 to 60, with higher scores indicating better self-efficacy. The questionnaire has shown excellent validity, reliability, and responsiveness in individuals with musculoskeletal disorders.
Social Support at Baseline | Baseline
  The French version of the Multidimensional Scale of Perceived Social Support (MSPSS) will be used to evaluate individual perceived satisfaction with social support received from family, friends and significant others. It is a 12 Likert-type items questionnaire with 7 response options (from 1, 'completely disagree', to 7 'strongly agree'). Higher scores represent higher satisfaction with social support received. The scale presented satisfactory internal consistency with a Cronbach's alpha value of 0.92.
Physical Activity Level at Baseline | Baseline
  The French short version of the International Physical Activity Questionnaire (IPAQ) will be used to assesses the frequency, duration, and intensity of physical activity. This short version includes 7 items and provides total activity scores expressed in metabolic equivalent (MET) minutes. A test-retest reliability of 0.81 (95% Confidence Interval 0.79 to 0.82) were previously determined.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Roy, PT, PhD, Principal Investigator — Laval University
Locations (1):
- Dayana P Rosa, Québec, Quebec, Canada